CLINICAL TRIAL: NCT05809063
Title: Characterization, Risk Factors and Outcome of Neonates Admitted to Neonatal Intensive Care Units (NICU) at Sohag University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rofida Abdelsabor Abdelbasset, Resident of pediatric and neonatology department, Sohag University Hospitals, Sohag University
Other Study IDs: Soh-Med-23-03-15MS
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Neonatal Diseases
MeSH Terms: conditions — Infant, Newborn, Diseases | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- cardiovascular patients: neonates that have cardiovascular diseases
  Interventions: Other: observational
- respiratory patients: neonates that have respiratory diseases
  Interventions: Other: observational
- gastrointestinal diseases: neonates that havegastrointestinal diseases
  Interventions: Other: observational
- renal patients: neonates that have renal diseases
  Interventions: Other: observational
- central nervous system diseases: neonates that have central nervous system diseases
  Interventions: Other: observational
- metabolic patients: neonates that have metabolic diseases
  Interventions: Other: observational
- endocrinal patients: neonates that have endocrinal diseases
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — document the number , disease pattern& outcome of neonates admitted to the neonatal intensive care units

SUMMARY:
The neonatal period considered the time from birth up to the first 28 days of life & further classified into:

* Very early birth (birth to < 24 hours).
* Early birth (24 hours to < 7 days).
* Late or last neonatal period (7 days to 28 days).

It is characterized by the transition from extra uterine life and rapid growth and development. It is the common vulnerable time or period of human life as it accounts for more high mortalities and morbidities, however, most of them are preventable.

The pattern of neonatal disease is a useful indicator of the availability, utilization and effectiveness of maternal and child health care services.

It varies from place to place and from time to time even in the same locality. Information on admission and mortality patterns of hospitalized neonates should reflect the major causes of illnesses and standard of care provided to neonates in a particular locality.

To improve neonatal services with better overall outcomes and less sever morbidities early identification of the risk factors is paramount so that appropriate interventions can be directed towards the most prevalent and treatable neonatal illnesses. To achieve this goal, it is important to study the pattern of neonatal admissions

ELIGIBILITY:
Inclusion Criteria:

* All neonates that will be admitted in Neonatal Intensive Care Units (NICU) including preterm, term and post term neonates.

Exclusion Criteria:

* Failure to obtain consent.
* Neonates need preparation for advanced interventions not available in our unit like cardiac operations.
* Neonates require peritoneal dialysis.
* Traumatic injury.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - All neonates that will be admitted in Neonatal Intensive Care Units (NICU) including preterm, term and post term neonates.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
document the number, & outcome in neonates with respiratory diseases admitted to neonatal intensive care units | 12 months
  all neonates admitted with respiratory diseases in neonatal intensive care units
document the number, & outcome in neonates with cardiovascular diseases admitted to neonatal intensive care units | 12 months
  all neonates admitted with cardiovascular diseases in neonatal intensive care units
document the number, & outcome in neonates with gastrointestinal diseases admitted to neonatal intensive care units | 12 months
  all neonates admitted with gastrointestinal diseases in neonatal intensive care units
document the number, & outcome in neonates with renal diseases admitted to neonatal intensive care units | 12 months
  all neonates admitted with renal diseases in neonatal intensive care units
document the number, & outcome in neonates with central nervous system diseases admitted to neonatal intensive care units | 12 months
  all neonates admitted with central nervous system diseases in neonatal intensive care units
document the number, & outcome in neonates with metabolic diseases admitted to neonatal intensive care units | 12 months
  all neonates admitted with metabolic diseases in neonatal intensive care units
document the number, & outcome in neonates with endocrinal diseases admitted to neonatal intensive care units | 12 months
  all neonates admitted with endocrinal diseases in neonatal intensive care units

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University hospitals, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Persson M, Shah PS, Rusconi F, Reichman B, Modi N, Kusuda S, Lehtonen L, Hakansson S, Yang J, Isayama T, Beltempo M, Lee S, Norman M; International Network for Evaluating Outcomes of Neonates. Association of Maternal Diabetes With Neonatal Outcomes of Very Preterm and Very Low-Birth-Weight Infants: An International Cohort Study. JAMA Pediatr. 2018 Sep 1;172(9):867-875. doi: 10.1001/jamapediatrics.2018.1811. PMID 29971428
- [Background] Mansoor KP, Ravikiran SR, Kulkarni V, Baliga K, Rao S, Bhat KG, Baliga BS, Kamath N. Modified Sick Neonatal Score (MSNS): A Novel Neonatal Disease Severity Scoring System for Resource-Limited Settings. Crit Care Res Pract. 2019 May 9;2019:9059073. doi: 10.1155/2019/9059073. eCollection 2019. PMID 31210987
- [Background] Dorling JS, Field DJ, Manktelow B. Neonatal disease severity scoring systems. Arch Dis Child Fetal Neonatal Ed. 2005 Jan;90(1):F11-6. doi: 10.1136/adc.2003.048488. PMID 15613564